CLINICAL TRIAL: NCT02127749
Title: The Role of the Gut Microbiota in the Systemic Immune Response During Human Endotoxemia
Acronym: MISSION-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, W.J. Wiersinga, MD, PhD, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NL45198.018.13; NL45198.018.13 (Other: CCMO (Centrale Commissie voor Mensgebonden Onderzoek))
Record Dates: First submitted 2014-04-28; First posted 2014-05-01 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Endotoxemia
Keywords: antibiotics; gut microbiota; endotoxemia; innate immunity
MeSH Terms: conditions — Endotoxemia | interventions — Endotoxins; Vancomycin; Metronidazole; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Experimental): Subjects are not pretreated with antibiotics Subjects receive 2 ng/kg endotoxin intravenously
  Interventions: Drug: Endotoxin
- Antibiotics (Experimental): Subjects are pretreated with broad-spectrum antibiotics: Vancomycin, Metronidazole, Ciprofloxacin Subjects receive 2 ng/kg endotoxin intravenously
  Interventions: Drug: Endotoxin; Drug: Vancomycin, Metronidazole, Ciprofloxacin

INTERVENTIONS:
Drug: Endotoxin — Both groups will receive 2 ng/kg LPS (endotoxin) intravenously
  Other Names: LPS
Drug: Vancomycin, Metronidazole, Ciprofloxacin — ciprofloxacin 500mg 2 times per day, vancomycin 500mg 3 times per day metronidazole 500mg 3 times per day All together during 7 days
  Arms: Antibiotics

SUMMARY:
The purpose of this study is to determine whether treatment with antibiotics, which harm the gut flora, causes the immune system to be less effective.

DETAILED DESCRIPTION:
Rationale: Sepsis ranks among the top ten leading causes of death worldwide. Most nonsurvivors die in a state of immunosuppression. The gut microbiota exerts numerous beneficial functions in the host response against infections. Gut flora components express microorganism-associated molecular patterns (MAMPs) such as lipopolysaccharide (LPS), which are recognized by pattern recognition receptors (PRRs) expressed by neutrophils and macrophages. MAMPs from the intestinal microbiota constitutively translocate to the circulation and prime bone marrow derived neutrophils via PRRs. Antibiotic treatment, which is standard of care for all patients with sepsis, depletes the gut microbiota and leads to a diminished release of MAMPs and other bacteria derived products. This causes diminished priming of systemic immunity, which may attribute to sepsis associated immunosuppression and an increased susceptibility to invading bacteria.

Objective: To investigate the role of the gut microbiota in the systemic priming of immune effector cells during human endotoxemia

Study design: Randomized, between- and within-subject-controlled intervention study in human volunteers

Intervention: All subjects will receive lipopolysaccharide (endotoxin; 2 ng/kg bodyweight) intravenously to induce experimental endotoxemia. Eight subjects will be pretreated with broad spectrum antibiotics (ciprofloxacin, vancomycin, metronidazole) for seven days (washout period of 36 hours before endotoxemia), in order to deplete the gut microbiota. Blood and faeces will be sampled before, during and after endotoxemia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male between 18 and 35 years of age
* Capable of giving written informed consent
* Chemistry panel without any clinically relevant abnormality
* Normal defecation pattern

Exclusion Criteria:

* Major illness in the past 3 months or any chronic medical illness
* History of any type of malignancy
* Past or current gastrointestinal disease
* Known positive test for hepatitis C antibody, hepatitis B surface antigen or HIV antibody 1 or 2
* Current or chronic history of liver disease
* Subject uses tobacco products
* History, within 3 years, of drug abuse
* History of alcoholism
* Any clinically relevant abnormality on the 12-lead ECG
* The subject has received an investigational product within three months
* Use of prescription or non-prescription drugs
* Use of antibiotics within 12 months
* Known allergy to antibiotics
* Subject has difficultly in donating blood or accessibility of a vein in left or right arm.
* Subject has donated more than 350 mL of blood in last 3 months
* Difficulty swallowing pills
* Body mass index more than 28

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cytokine production in blood | within 8 hours after LPS administration

CONTACTS AND LOCATIONS:
Overall Officials: W. J. Wiersinga, MD, PhD, Principal Investigator — Academic Medical Centre, Amsterdam
Locations (1):
- Academic Medical Centre, Amsterdam, Netherlands

REFERENCES:
- [Derived] Haak BW, Lankelma JM, Hugenholtz F, Belzer C, de Vos WM, Wiersinga WJ. Long-term impact of oral vancomycin, ciprofloxacin and metronidazole on the gut microbiota in healthy humans. J Antimicrob Chemother. 2019 Mar 1;74(3):782-786. doi: 10.1093/jac/dky471. PMID 30418539
- [Derived] Lankelma JM, Cranendonk DR, Belzer C, de Vos AF, de Vos WM, van der Poll T, Wiersinga WJ. Antibiotic-induced gut microbiota disruption during human endotoxemia: a randomised controlled study. Gut. 2017 Sep;66(9):1623-1630. doi: 10.1136/gutjnl-2016-312132. Epub 2016 Jun 15. PMID 27307305